CLINICAL TRIAL: NCT01190696
Title: Study of Surgical Method Versus Casting for Treatment of Femoral Fracture in Children
Brief Title: Titanium Elastic Nailing Versus Hip Spica Cast in Treatment of Femoral Fractures in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Dr. Alireza Yousefy/Associate Professor of Medical Education, Isfahan University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASD-1213-5
Record Dates: First submitted 2010-08-27; First posted 2010-08-30 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2009-02

CONDITIONS: Femoral Shaft Fracture
Keywords: Spica Cast; TEN; Femoral Shaft Fracture; Children

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hip spica casting (Other): Patients in the spica cast group treated with skeletal traction and spica cast applied for them
  Interventions: Device: Hip spica casting
- titanium elasting nailing (Other): For patients in the Titanium Elasting Nailing group, the nail applied retrogradely in femoral shaft fracture
  Interventions: Procedure: titanium elastic nailing

INTERVENTIONS:
Procedure: titanium elastic nailing — we inserted titanium nail in femoral fractures retrogradely
  Other Names: TEN
  Arms: titanium elasting nailing
Device: Hip spica casting — we applied cast for three weeks in patients with femoral shaft fracture
  Other Names: TEN
  Arms: hip spica casting

SUMMARY:
The purpose of this study is to determine which method is better for treatment of femoral fracture in children in outcomes.

DETAILED DESCRIPTION:
There is no consensus on treatment of closed femoral shaft fractures in children 6-12years old. We aimed to compare hip spica cast with titanium elastic nailing (TEN) in the treatment of femoral shaft fractures in children.

ELIGIBILITY:
Inclusion Criteria:

* patients 6-12 years old with femoral shaft fracture without exclusion criteria

Exclusion Criteria:

* Segmental, Winquist type III and IV comminuted fractures, previously diagnosed neuromuscular disease (e.g., cerebral palsy), metabolic bone disorders (e.g. osteomalacia), or pathological fractures.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | at 1 months post-operatively
  identification of Length of hospital stay (days)for patients who treated with titanium elastic nailing or casting

SECONDARY OUTCOMES:
the time to walking with aids | at 1 months post-operatively
  identification of the time to walking with aids in patients who treated with titanium elastic nailing or casting
parent's satisfaction | at 1 months post-operatively
  identification of parent's satisfaction with questionnair in patients who treated with titanium elastic nailing or casting
the time absent from school | at 1 months post-operatively
  identification of the time absent from school in patients who treated with titanium elasting nailing or casting

CONTACTS AND LOCATIONS:
Overall Officials: hamidreza shemshaki, MD, Study Chair — MD,research comittee
Locations (1):
- Al-zahra university hospital, Isfahan, Isfahan, Iran